CLINICAL TRIAL: NCT01780428
Title: A Double-Blind, Randomized, Placebo-Controlled, Multiple-dose Multi-Center Phase III Study of the Safety and Efficacy of Cl-108 in the Treatment of Moderate to Severe Pain
Brief Title: Phase III Study of the Safety and Efficacy of Cl-108 in the Treatment of Moderate to Severe Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charleston Laboratories, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: CLCT-002
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Pain; Nausea; Vomiting
Keywords: Pain; Nausea; Vomiting
MeSH Terms: conditions — Pain; Nausea; Vomiting | interventions — Acetaminophen; Promethazine; oxycodone-acetaminophen; Hydrocodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- CL-108 (Experimental): CL-108 (hydrocodone 7.5 mg, acetaminophen 325 mg, Promethazine 12.5 mg)
  Interventions: Drug: CL-108 (hydrodocone 7.5 mg, acetaminophen 325 mg, promethazine 12.5 mg)
- Norco (Active Comparator): Commercial product containing hydrocodone 7.5 mg. acetaminophen 325 mg
  Interventions: Drug: CL-108 (hydrodocone 7.5 mg, acetaminophen 325 mg, promethazine 12.5 mg)
- Placebo (Placebo Comparator): CL-108 formulation without API
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CL-108 (hydrodocone 7.5 mg, acetaminophen 325 mg, promethazine 12.5 mg)
  Other Names: Norco (hydrocodone 7.5 mg, acetaminophen 325 mg); Placebo
  Arms: CL-108; Norco
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, multiple-dose, placebo- and positive-controlled study of CL-108 (hydrocodone 7.5 mg/APAP 325 mg, promethazine 12.5 mg) in patients with moderate to severe pain following surgical removal of impacted third molar teeth.

A positive control ( Norco, a commercial formulation of hydrocodone 7.5 mg/APAP 325 mg) was included to determine the anti-emetic effects of CL-108. The efficacy of CL-108 was also evaluated to placebo for the relief of pain.

ELIGIBILITY:
Inclusion Criteria:

* Determination of being likely or possibly nausea-prone.
* Male or non-pregnant and non-lactating female.
* Surgical extraction of at least 2 impacted third molar teeth
* A female of child-bearing potential is eligible to participate in this study if she has a negative urine pregnancy test and is using an acceptable method of birth control.
* Surgical extraction of at least 2 impacted third molar teeth.
* Presence of at least moderate post-operative pain.

Exclusion Criteria:

* Medial Condition, presence of a serious medical condition.
* Active local infection.
* Drug Allergy history of hypersensitivity to an Opioid, Promethazine, Acetaminophen.
* Caffeine use since midnight before the operation.
* Use of an IND Drug within past 30 days.
* Previous participation in this study.
* Pregnant or lactating.
* Employee of the PI,sub-investigator or Charleston Labs or relative of an employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To compare the occurrence and severity of opioid-induced nausea and vomiting (OINV) associated with CL-108 to Norco. | Over the first 24 hours
  After data has been locked.
To demonstrate the efficacy of CL-108 when compared to placebo for the relief of pain following surgical removal of impacted third molar teeth. | over 24 hours (SPID24)
  After data has been locked.

SECONDARY OUTCOMES:
Reduction of the severity of nausea in patients treated with an opioid-containing pain reliever. | over 6 hours
  After data lock.
Reduction of vomiting in patients treated with an opioid-containing pain reliever. | over 6 hours
  After data lock.

OTHER OUTCOMES:
Elimination of vomiting in patients treated with an opioid-containing pain reliever. | 6 hours and 24 hours
  After data lock.
Elimination of nausea in patients treated with an opioid-containing pain reliever. | 6 hours and 24 hours
  After data lock.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Charleston Website — http://www.charlestonlabs.com